CLINICAL TRIAL: NCT02059278
Title: A Randomized, Multicenter, Parallel-Group, Observer-Masked, Phase 3 Study to Compare the Safety and Efficacy of T-2345 Ophthalmic Solution to Xalatan (Latanoprost 0.005%) in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: Safety and Efficacy of T-2345 Compared to Xalatan in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nephron Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T-2345-001
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2017-12

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Primary open angle glaucoma; Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- T-2345 (Experimental): T-2345 Ophthalmic Solution dosed 1 drop QD in the eye(s) in the evening (8 pm +/- 30 minutes)
  Interventions: Drug: T-2345
- Xalatan (Experimental): Xalatan (Latanoprost 0.005% Ophthalmic Solution) dosed 1 drop QD in the eye(s) in the evening (8 pm +/- 30 minutes)
  Interventions: Drug: Xalatan

INTERVENTIONS:
Drug: T-2345 — T-2345 Ophthalmic Solution
  Arms: T-2345
Drug: Xalatan — Xalatan (latanoprost 0.005% ophthalmic solution)
  Arms: Xalatan

SUMMARY:
This is a Phase 3 study to evaluate the safety and efficacy of T-2345 dosed to one of both eyes once daily for 84 days compared to Xalatan dosed to one of both eyes once daily for 84 days in patients with elevated eye pressure.

DETAILED DESCRIPTION:
The objective of this Phase 3 study is to evaluate the efficacy and safety of T-2345 nonpreserved ophthalmic solution (latanoprost 0.005%) in comparison to Xalatan® (latanoprost 0.005%) in subjects with primary open angle glaucoma (POAG) or ocular hypertension (OH).

This will be a randomized, multicenter, parallel-group, observer-masked study in approximately 380 evaluable subjects treated for 84 days. Subjects will have a history of POAG or OH and elevated intraocular pressure (IOP) and will have been adequately controlled (IOP ≤ 18 mm Hg) on latanoprost 0.005% ophthalmic solution monotherapy for at least 4 weeks.

Primary efficacy (IOP) will be assessed in the study eye at each visit by Goldmann applanation tonometry at all assessment visits.

Safety will be assessed at each visit by corrected Snellen Visual Acuity, slit lamp examination/anterior chamber cell count and flare and adverse event (AE) collection.

Primary Efficacy Endpoint is the between-group comparison of the mean IOP values at each time point at each of the Day 15, 42, and 84 visits.

Secondary Efficacy Endpoints include:

* Between-group comparison of the mean change from baseline in diurnal IOP measurements at all postbaseline visits.
* Between-group comparison of the mean change from baseline in IOP measurements at all times points at Day 15, Day 42 and Day 84.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. POAG or OH with IOP treated and adequately controlled (IOP ≤ 18 mm Hg) with latanoprost 0.005% ophthalmic solution monotherapy for at least 4 weeks prior to Screening.
3. Each eye being treated with latanoprost 0.005% ophthalmic solution monotherapy must have mean IOP ≤ 18 mm Hg at Screening and mean IOP ≤ 28 mm Hg at Baseline; measurements will be taken at each visit at 8 AM, 10 AM, and 4 PM (each ± 30 minutes) with AM measurements of IOP at least 2 hours apart. If only one eye qualifies but both eyes have glaucoma and the fellow eye will require antiglaucoma medications, the subject does not qualify for the trial.
4. Stable visual field (VF), defined as no sign of VF degradation between two consecutive 30-2 or two consecutive 24-2 VF examinations. For subjects with no VF defect (eg, those with OH), a single, normal VF examination performed ˂ 6 months prior to the screening visit is allowed to determine eligibility. For patients who have an abnormal VF examination, the following criteria apply:

   * Two VF (most recent VF and past VF) examinations performed at least ≥ 6 months and ≤ 18 months apart must be compared;
   * The most recent VF examination should be performed < 6 months prior to the Screening visit;
   * The past VF examination should be performed ≥ 6 months and ≤ 18 months prior to the most recent VF test.
5. Stable corrected Snellen visual acuity (VA) of better than 20/200 in the study eye. Patients must see ≥ 50% of the letters on a single line to accept that VA line.
6. Central corneal thickness 480-620 μm in the study eye.
7. Shaffer gonioscopic grade of ≥ 3 (in at least 3 quadrants) in both eyes.
8. Female subjects must be 1-year postmenopausal, surgically sterilized, or women of childbearing potential with a negative urine pregnancy test at Screening. Women of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include the use of at least one of the following: intrauterine (intrauterine device), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.
9. All subjects must provide signed written consent prior to participation in any study-related procedures.

Exclusion Criteria:

In the study eye:

1. A mean deviation of < -20 dB on VF examination.
2. A mean IOP ˃ 28 mm Hg at Baseline.
3. Presence of a scotoma within 5° of fixation on VF examination.
4. Aphakia.
5. Use of any antiglaucoma medication in addition to latanoprost 0.005% ophthalmic solution within 2 weeks prior to Screening and any antiglaucoma medication (other than latanoprost) during the study period other than the randomized study medication.
6. Use of any topical ophthalmic steroid within 2 weeks prior to Baseline. A short course of oral steroids is acceptable if the course is completed > 2 weeks prior to Screening. Inhaled and intranasal steroids are acceptable.
7. Use of topical nonsteroidal anti-inflammatory drug (NSAID) within 2 weeks prior to Baseline.
8. Use of any ophthalmic medications during the study period (nonpreserved artificial tears are allowed).
9. Ocular surgery or laser treatment of any kind in the study eye within 3 months prior to Baseline.
10. History of ocular allergy/inflammation and/or severe blepharitis and/or uveitis. Seasonal allergic conjunctivitis is acceptable (avoid enrollment of subjects who may experience seasonal flare-up during the study period). Mild blepharitis/blepharoconjunctivitis, typically associated with prostaglandin usage, on the lid is acceptable.
11. History of ocular trauma or ocular infection within 3 months of Screening.
12. History of herpes simplex keratitis.
13. Current proliferative diabetic retinopathy or age-related macular degeneration, unless deemed not clinically significant by the Investigator.
14. Severe dry eye (eg, clinically relevant superficial punctate keratitis, epithelial erosions of the cornea, and/or use of dry eye medication [including artificial tears] with a frequency exceeding 8 instillations per day).
15. Contact lens wear during the study period. Contact lens wear in an untreated fellow eye is allowed.
16. Any secondary glaucoma or OH (eg, congenital glaucoma, closed-angle glaucoma, uveitic glaucoma, or pseudoexfoliation syndrome).
17. Any severe glaucoma defined by cupping (cup-to-disc ratio ≥ 0.8).
18. Any non-laser glaucoma surgery.
19. Any abnormality preventing accurate assessment (eg, resulting in unreliable applanation tonometry or VF examination).

    General:
20. Pregnancy or lactation.
21. Uncontrolled asthma (defined as asthma that does not respond to the maximum guideline-directed therapy).
22. Allergy to benzalkonium chloride.
23. History of moderate or severe renal or hepatic impairment.
24. Participation in any study of an investigational product within 30 days prior to Screening or at any time during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- El Paso, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T-2345 | Xalatan
Started | 165 | 170
Completed | 162 | 166
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Ran out of IP and decided to discontinue | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | T-2345 | Xalatan | Total
Number analyzed (Participants) | 164 | 170 | 334
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (10.2) | 66.1 (11.0) | 66.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 100 | 204
  Male | 60 | 70 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 22 | 40
  Not Hispanic or Latino | 146 | 148 | 294
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 28 | 65
  White | 125 | 141 | 266
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 164 | 170 | 334
Corneal thickness, study eye (μm) [Mean (Standard Deviation); unit: μm] | 550.7 (33.9) | 548.7 (34.5) | 549.6 (34.2)
Corneal thickness, fellow eye (μm) [Mean (Standard Deviation); unit: μm] | 552.1 (33.7) | 549.4 (33.6) | 550.7 (33.6)
Shaffer angle by gonioscopy, study eye [Count of Participants; unit: Participants] — Shaffer Angle is a measure of the anterior chamber angle based on a scale from 0 (closed) to IV (wide open). Shaffer Angles Grade III and IV are considered to be angles where closure is not possible and normal drainage can occur to reduce intraocular pressure.
  Participants
    Schaffer Angle Grade III | 83 | 84 | 167
    Schaffer Angle Grade IV | 81 | 86 | 167
Shaffer angle by gonioscopy, fellow eye [Count of Participants; unit: Participants] — Shaffer Angle is a measure of the anterior chamber angle based on a scale from 0 (closed) to IV (wide open). Shaffer Angles Grade III and IV are considered to be angles where closure is not possible and normal drainage can occur to reduce intraocular pressure.
  Participants
    Schaffer Angle Grade III | 83 | 84 | 167
    Schaffer Angle Grade IV | 81 | 86 | 167

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: Evaluation of intraocular pressure using Goldmann applanation tonometry.
  Primary outcome was the between group difference in the change from baseline in IOP at each of 9 assessment points.
  Equivalence was achieved if the 95% Confidence Intervals were within 1.5 mmHg at all 9 time points
Time Frame: Measured at 8am 10 am and 4 pm at Baseline and on Days 15, 42 and 84
Population: The Per Protocol population was the primary efficacy population and consisted of those subjects in the ITT population who had no major protocol violations and no missing data points
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | T-2345 | Xalatan
Number analyzed (Participants) | 161 | 164
mm Hg
  Day 15 08:00 | -3.0 (3.2) | -3.8 (3.4)
  Day 15 10:00 | -2.7 (2.9) | -3.6 (3.3)
  Day 15 16:00 | -2.3 (2.8) | -3.1 (3.3)
  Day 42 08:00 | -3.0 (3.2) | -3.5 (3.2)
  Day 42 10:00 | -2.7 (3.1) | -3.5 (3.4)
  Day 42 16:00 | -2.3 (2.9) | -3.1 (3.4)
  Day 84 08:00 | -3.0 (3.2) | -3.5 (3.2)
  Day 84 10:00 | -2.7 (3.0) | -3.6 (3.1)
  Day 84 16:00 | -2.2 (2.8) | -2.9 (3.2)
Statistical Analysis 1: Comparison: T-2345 vs Xalatan; The primary endpoint was measured at 9 separate assessment times (3 time points over a 12 hour period on 3 separate days. The primary analysis was based on a comparison of the IOP change from baseline between the two arms at each assessment.The equivalence margin was tested using an analysis of covariance on change from baseline with pooled site and baseline as a factor. Equivalence was considered to be met if the 95% confidence intervals were within 1.5 mmHg at each of the 9 assessment points; Test type: Equivalence — Analysis at 8 am on Day 15; p = 0.0091, ANCOVA; Mean Difference (Final Values) = 0.781, 95% CI 2-sided [0.195 to 1.366] — ANCOVA on change from baseline at 8 am on Day 15
Statistical Analysis 2: Comparison: T-2345 vs Xalatan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Analysis at 10 am on Day 15; p = 0.0098, ANCOVA; Mean Difference (Final Values) = 0.664, 95% CI 2-sided [0.161 to 1.167] — ANCOVA on change from baseline at 10 am on Day 15
Statistical Analysis 3: Comparison: T-2345 vs Xalatan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Analysis at 4 pm on Day 15; p = 0.0398, ANCOVA; Mean Difference (Final Values) = 0.542, 95% CI 2-sided [0.025 to 1.058] — ANCOVA on change from baseline at 4 pm on Day 15
Statistical Analysis 4: Comparison: T-2345 vs Xalatan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Analysis at 8 am on Day 42; p = 0.1008, ANCOVA; Mean Difference (Final Values) = 0.478, 95% CI 2-sided [-0.093 to 1.050] — ANCOVA on change from baseline at 8 am on Day 42
Statistical Analysis 5: Comparison: T-2345 vs Xalatan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Analysis at 10 am on Day 42; p = 0.0558, ANCOVA; Mean Difference (Final Values) = 0.505, 95% CI 2-sided [-0.013 to 1.024] — ANCOVA on change from baseline at 10 am on Day 42
Statistical Analysis 6: Comparison: T-2345 vs Xalatan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Analysis at 4 pm on Day 42; p = 0.0491, ANCOVA; Mean Difference (Final Values) = 0.538, 95% CI 2-sided [0.002 to 1.074] — ANCOVA on change from baseline at 4 pm on Day 42
Statistical Analysis 7: Comparison: T-2345 vs Xalatan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Analysis at 8 am on Day 84; p = 0.0025, ANCOVA; Mean Difference (Final Values) = 0.808, 95% CI 2-sided [0.286 to 1.329] — ANCOVA on change from baseline at 8 am on Day 84
Statistical Analysis 8: Comparison: T-2345 vs Xalatan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Analysis at 10 am on Day 84; p = 0.0113, ANCOVA; Mean Difference (Final Values) = 0.627, 95% CI 2-sided [0.143 to 1.111] — ANCOVA on change from baseline at 10 am on Day 84
Statistical Analysis 9: Comparison: T-2345 vs Xalatan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Analysis at 4 pm on Day 84; p = 0.0649, ANCOVA; Mean Difference (Final Values) = 0.456, 95% CI 2-sided [-0.063 to 0.975] — ANCOVA on change from baseline at 4 pm on Day 84

2. Secondary Outcome: Visual Acuity
Description: Visual Acuity was measured using the Corrected Snellen Visual Acuity method reported as the Logarithm Minimum Angle of Resoution (logMAR) change from baseline. The Snellen eye chart was used with the subject's current corrected lens prescription at a distance equivalent to 20 feet. Results from the Snellen chart were converted to the logMAR scale which is the standard tool for reporting visual acuity outcomes.
Time Frame: Baseline and 84 days
Population: Safety population defined as all randomized subjects who received at least one dose of the allocated study medication.
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | T-2345 | Xalatan
Number analyzed (Participants) | 165 | 169
logMAR units | -0.003 (0.075) | -0.008 (0.082)

3. Secondary Outcome: Slit Lamp Examination
Description: Number of participants with eye abnormalities following routine slit lamp examination. The anterior segment of the eye including lids, cornea, conjunctiva, anterior chamber, iris and lens were evaluated with a routine slit lamp examination and any abnormalities observed were reported.
Time Frame: Baseline and 84 days
Population: Safety population defined as all randomized subjects who received at least one dose of the allocated study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | T-2345 | Xalatan
Number analyzed (Participants) | 165 | 169
Participants
  Lid | 4 | 0
  Cornea | 1 | 2
  Conjunctiva | 2 | 2
  Iris | 0 | 1
  Lens | 3 | 6

4. Secondary Outcome: Ophthalmoscopy
Description: Number of participants with eye abnormalities following ophthalmoscopy. Direct ophthalmoscopy with dilation included assessment of the optic nerve head for pallor and cupping. A dilated fundus examination consisting of the vitreous, optic nerve, macula, and peripheral retina was conducted. Results are reported as the number of subjects with clinical significant abnormalities at Day 84 that were not clinically significant at Baseline.
Time Frame: Baseline and 84 days
Population: Safety population defined as all randomized subjects who received at least one dose of the allocated study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | T-2345 | Xalatan
Number analyzed (Participants) | 165 | 169
Participants
  Study eye | 1 | 0
  Fellow eye | 1 | 0

5. Secondary Outcome: Mean Deviation in Visual Field
Description: Visual Field was performed using an automated perimeter according to the sites standard protocol. This test measures the angle of the visual field from the central visual axis. Visual Field Testing generates a numerical scale as its main result which shows the retinal sensitivities at the different test locations, expressed in Decibels (dB). The mean deviation in the visual field reflects the overall depression (deviation from normal values). Negative values indicate a reduction in visual field. The analysis performed is the mean change from baseline at Day 84.
Time Frame: Baseline and 84 days
Population: Safety population defined as all randomized subjects who received at least one dose of the allocated study medication.
Measure: Mean (Standard Deviation); unit: Decibels (dB)
Arm/Group | T-2345 | Xalatan
Number analyzed (Participants) | 165 | 169
Decibels (dB)
  Study eye | -0.169 (1.607) | -0.166 (1.680)
  Fellow eye | 0.067 (2.124) | -0.094 (1.466)

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | T-2345 | Xalatan
All-Cause Mortality (participants affected / at risk) | 0/165 | 1/169
Serious Adverse Events (participants affected / at risk) | 1/165 | 4/169
Other Adverse Events (participants affected / at risk) | 23/165 | 44/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-2345 (N=165) | Xalatan (N=169)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal ganglia stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-2345 (N=165) | Xalatan (N=169)
Conjunctival hyperemia (Eye disorders) | 3 (3) | 4 (4)
Blepharitis (Eye disorders) | 2 (2) | 5 (5)
Punctate keratitis (Eye disorders) | 1 (1) | 5 (5)
Vitreous detachment (Eye disorders) | 1 (1) | 2 (2)
Conjunctival cyst (Eye disorders) | 0 (0) | 2 (2)
Conjunctival hemorrhage (Eye disorders) | 0 (0) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 2 (2)
Instillation site pain (General disorders) | 3 (3) | 8 (8)
Instillation site pruritus (General disorders) | 2 (2) | 1 (1)
Instillation site abnormal sensation (General disorders) | 1 (1) | 2 (2)
instillation site complication (General disorders) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Sciatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes